CLINICAL TRIAL: NCT00277212
Title: A Multicenter, Double-blind, Study of the Efficacy and Safety of Aripiprazole in Combination With Lamotrigine in the Long-term Maintenance Treatment of Patients With Bipolar I Disorder With a Recent Manic or Mixed Episode
Brief Title: A Phase IV Study of the Safety and Efficacy of Aripiprazole in Combination With Lamotrigine in the Long-Term Maintenance Treatment of Patients With Bipolar I Disorder With A Recent Manic or Mixed Episode
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN138-392 ST
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Results first posted 2010-10-20 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder with a recent manic or mixed episode
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Experimental): Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole ; Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
  Interventions: Drug: Lamotrigine + Aripiprazole
- A2 (Placebo Comparator): Phase 2 Double-Blind Treatment: Lamotrigine + Placebo
  Interventions: Drug: Lamotrigine + Placebo

INTERVENTIONS:
Drug: Lamotrigine + Aripiprazole — Tablets, Oral, once daily, Phase 1 (all subjects) - up to 24 weeks; Phase 2 - up to 52 weeks
  Lamotrigine 100-200 mg/day
  Aripiprazole 10-30 mg/day
  Other Names: Abilify; BMS-337039
  Arms: A1
Drug: Lamotrigine + Placebo — Tablets, Oral, once daily, Phase 2 - up to 52 weeks
  Lamotrigine 100-200 mg/day
  placebo 0 mg/day
  Arms: A2

SUMMARY:
Efficacy of Aripiprazole in Combination with Lamotrigine in the Long-Term Maintenance Treatment of Bipolar I Disorder in Outpatients with Recent Manic or Mixed Episode

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (Text Revision) (DSM-IV-TR) criteria for bipolar I disorder, recently experiencing a manic or mixed episode with a history of one or more manic or mixed episodes of sufficient severity to require treatment with a mood stabilizer or antipsychotic

Exclusion Criteria:

* First manic episode
* Current manic or mixed episode with > 2 years duration
* Treated with aripiprazole within the past 3 months
* Allergic, intolerant, hypersensitive or refractory to aripiprazole or lamotrigine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1169 (Actual)
Dates: Start 2005-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (66):
- United States (62):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Southwest Biomedical Research Foundation, Tucson, Arizona
  - Pravin Kansagra, M.D., Anaheim, California
  - College Hospital Costa Mesa, Costa Mesa, California
  - Pacific Institute For Medical Research, Inc., Los Angeles, California
  - Excell Research, Oceanside, California
  - Southern Ca Clinical Research, Inc., Pasadena, California
  - Stanford University, Stanford, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Health Sciences America, Llc, Boca Raton, Florida
  - Cns Clinical Research Group, Coral Springs, Florida
  - Act Clinical Research Institute, Llc, Daytona Beach, Florida
  - Neuropsychiatric Research Center Of Southwest Florida, Fort Myers, Florida
  - Aurora-Cuervo Clinical Trials, Miami, Florida
  - Gulf Coast Medical Research, Port Charlotte, Florida
  - Janus Center For Psychiatric Research, West Palm Beach, Florida
  - Comprehensive Neuroscience, Inc, Atlanta, Georgia
  - Valle Vista Health System, Greenwood, Indiana
  - Clinco, Terre Haute, Indiana
  - Clinical Trials Technology, Inc, Prairie Village, Kansas
  - Clinical Research Institute, Wichita, Kansas
  - University Of Kentucky, Dept. Of Psychiatry, Lexington, Kentucky
  - Owensboro Behavioral Care, Owensboro, Kentucky
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Clinical Insights, Glen Burnie, Maryland
  - Capital Clinical Research Associates, Rockville, Maryland
  - Psychopharmacology Research Corporation, Farmington Hills, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - University Of Medicine & Dentistry Of New Jersey, Cherry Hill, New Jersey
  - Buffalo Psychiatric Center, Buffalo, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Duke University Medical Center, Durham, North Carolina
  - Zarzar Psychiatric Associates, Pllc, Raleigh, North Carolina
  - Horizon Medical Services, Bismarck, North Dakota
  - Neuro Behavioral Clinical Research, Inc., Canton, Ohio
  - Community Research, Cincinnati, Ohio
  - Saroj Brar Md, Inc, Cleveland, Ohio
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Lehigh Center For Clinical Research, Allentown, Pennsylvania
  - Dubois Regional Medical Center, DuBois, Pennsylvania
  - Freimer, Martin, East Stroudsburg, Pennsylvania
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Belmont Center For Comprehensive Treatment, Philadelphia, Pennsylvania
  - Cns Research Institute, Philadelphia, Pennsylvania
  - Ut Medical Group/Odyssey Research, Memphis, Tennessee
  - Psychiatric Consultants, Pc, Nashville, Tennessee
  - Harmony Research, Llc, Piney Flats, Tennessee
  - Bayou City Research, Ltd., Houston, Texas
  - Alamo Superior Research, San Antonio, Texas
  - University Of Virginia Health System, Charlottesville, Virginia
  - Windwood Centre, Virginia Beach, Virginia
  - Pacific Institute Of Medical Sciences, Bothell, Washington
  - Summit Research Network (Seattle) Llc, Seattle, Washington
  - Health Research Center, Morgantown, West Virginia
  - Aurora Health Care, Milwaukee, Wisconsin
- Puerto Rico (4):
  - Local Institution, Cabo Rojo
  - Local Institution, Ponce
  - Local Institution, Rio Piedras
  - Local Institution, San Juan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1169 patients were enrolled in the study; 382 participants were considered baseline failures and did not enter Phase 1.
Groups:
- Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole: Lamotrigine 100-200 mg/day, Aripiprazole 10-30 mg/day: tablets, oral, once daily, Phase 1 (all subjects) - up to 24 weeks
- Phase 2 Double-Blind Treatment: Lamotrigine + Placebo: Lamotrigine 100-200 mg/day, Placebo 0 mg/day: tablets, oral, once daily, Phase 2 - up to 52 weeks
- Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole: Lamotrigine 100-200 mg/day, Aripiprazole 10-30 mg/day: tablets, oral, once daily, Phase 2 - up to 52 weeks.
Period: Phase 1 - Single-Blind Treatment
Arm/Group | Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Started | 787 | 0 | 0
Phase 1 Safety Sample | 787 | 0 | 0
Phase 1 Efficacy Sample | 756 | 0 | 0
Completed | 352 | 0 | 0
Not Completed | 435 | 0 | 0
Not completed — Lack of Efficacy | 61 | 0 | 0
Not completed — Adverse Event | 93 | 0 | 0
Not completed — Withdrawal by Subject | 96 | 0 | 0
Not completed — Lost to Follow-up | 87 | 0 | 0
Not completed — Poor/Noncompliance | 35 | 0 | 0
Not completed — Pregnancy | 6 | 0 | 0
Not completed — Subject No Longer Met Study Criteria | 44 | 0 | 0
Not completed — Administrative Reason by Sponsor | 1 | 0 | 0
Not completed — Other Reasons | 12 | 0 | 0
Period: Phase 2 - Double-Blind Treatment
Arm/Group | Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Started | 0 | 173 | 178 (1 participant did not want to continue in the study for personal reasons, and did not enter Phase 2.)
Phase 2 Safety Sample | 0 | 165 | 176
Phase 2 Efficacy Sample | 0 | 164 | 174
Completed | 0 | 53 | 65
Not Completed | 0 | 120 | 113
Not completed — Lack of Efficacy | 0 | 54 | 39
Not completed — Adverse Event | 0 | 10 | 16
Not completed — Withdrawal by Subject | 0 | 17 | 16
Not completed — Lost to Follow-up | 0 | 18 | 18
Not completed — Poor/Noncompliance | 0 | 7 | 8
Not completed — Pregnancy | 0 | 2 | 2
Not completed — Subject No Longer Meets Study Criteria | 0 | 4 | 6
Not completed — Administrative Reasons By Sponsor | 0 | 1 | 3
Not completed — Other reasons | 0 | 7 | 5

BASELINE CHARACTERISTICS:
Arm/Group | Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole
Number analyzed (Participants) | 796
Age Continuous [Mean (Standard Deviation); unit: years] | 38.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 505
  Male | 291
Race/Ethnicity, Customized [Number; unit: participants]
  White | 693
  Black/African American | 88
  Asian | 10
  American Indian/Alaska Native | 2
  Native Hawaiian/Other Pacific Islander | 1
  Other | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 93
  Not Hispanic or Latino | 703
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (7.6)
Weight [Mean (Standard Deviation); unit: kg] | 84.7 (22.7)
BMI Category [Number; unit: participants]
  18.5 <= BMI <25 | 221
  25 <= BMI <30 | 215
  BMI <18.5 | 12
  BMI >=30 | 321
  Missing | 27

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Not Experiencing Relapse Through Week 52 in the Double-Blind Relapse Assessment Phase (Phase 2)
Description: Time from randomization to relapse to a manic or mixed episode in the Double-Blind Relapse Assessment Phase as measured by the Proportion of Participants without Relapse Through Week 52 (Kaplan-Meier's estimated survival rate).
Time Frame: Weeks 0, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Randomized Participants (comprises all patients who are randomized in Phase 2). n= number of randomized participants evaluated at given time point.
Measure: Number; unit: Proportion of Participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 173 | 178
Proportion of Participants
  Week 0 (n=173, n=178) | 1.00 | 1.00
  Week 2 (n=162, n=172) | 0.98 | 0.98
  Week 4 (n=154, n=159) | 0.97 | 0.96
  Week 6 (n=142, n=147) | 0.95 | 0.93
  Week 8 (n=135, n=135) | 0.93 | 0.90
  Week 12 (n=121, n=127) | 0.89 | 0.90
  Week 16 (n=101, n=127) | 0.88 | 0.90
  Week 20 (n=94, n=127) | 0.88 | 0.90
  Week 24 (n=86, n=127) | 0.84 | 0.90
  Week 28 (n=79, n=127) | 0.81 | 0.90
  Week 32 (n=69, n=83) | 0.78 | 0.89
  Week 36 (n=67, n=83) | 0.78 | 0.89
  Week 40 (n=62, n=83) | 0.77 | 0.89
  Week 44 (n=62, n=83) | 0.77 | 0.89
  Week 48 (n=62, n=83) | 0.77 | 0.89
  Week 52 (n=62, n=83) | 0.77 | 0.89
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Test type: Superiority or Other; p = 0.058, Log Rank — stratified Log-Rank test, controlling for type of index mood episode; Cox Proportional Hazard = 0.552, 95% CI 2-sided [0.296 to 1.030] — Cox's proportional hazards model, with type of index modd episode as stratification factor, and randomized treatment group as covariate

2. Secondary Outcome: Proportion of Participants Not Experiencing Relapse (Manic, Mixed, Depressive) in the Double-blind Relapse Assessment Phase Phase 2
Description: Proportion of Participants without Relapse Through Week 52 (Kaplan-Meier's estimated survival rate).
Time Frame: Weeks 0, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 1
Measure: Number; unit: Proportion of Participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 173 | 178
Proportion of Participants
  Week 0 (n=173, n=178) | 1.00 | 1.00
  Week 2 (n=163, n=175) | 0.96 | 0.95
  Week 4 (n=154, n=160) | 0.91 | 0.91
  Week 6 (n=145, n=149) | 0.87 | 0.88
  Week 8 (n=135, n=136) | 0.83 | 0.84
  Week 12 (n=121, n=123) | 0.76 | 0.82
  Week 16 (n=102, n=113) | 0.75 | 0.80
  Week 20 (n=94, n=111) | 0.74 | 0.80
  Week 24 (n=91, n=95) | 0.69 | 0.78
  Week 28 (n=78, n=85) | 0.65 | 0.77
  Week 32 (n=69, n=83) | 0.62 | 0.75
  Week 36 (n=67, n=76) | 0.62 | 0.74
  Week 40 (n=62, n=70) | 0.61 | 0.73
  Week 44 (n=62, n=70) | 0.61 | 0.73
  Week 48 (n=62, n=70) | 0.61 | 0.73
  Week 52 (n=19, n=70) | 0.58 | 0.73
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Test type: Superiority or Other; p = 0.055, Log Rank — p-value for equality of survival curves; stratified log-rank test, controlling for type of index mood episode; Hazard Ratio (HR) = 0.671, 95% CI 2-sided [0.446 to 1.011] — aripiprazole/placebo; Cox's proportional hazards model, with type of index mood episode as stratification facto, and randomized treatment group as covariate

3. Secondary Outcome: Proportion of Participants Not Experiencing a Depressive Relapse in the Double-blind Relapse Assessment Phase (Phase 2)
Description: Proportion of Participants without Relapse Through Week 52 (Kaplan-Meier's estimated survival rate).
Time Frame: Weeks 0, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 1
Measure: Number; unit: Proportion of Participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 173 | 178
Proportion of Participants
  Week 0 (n=173, n=178) | 1.00 | 1.00
  Week 2 (n=163, n=175) | 0.98 | 0.98
  Week 4 (n=151, n=160) | 0.94 | 0.95
  Week 6 (n=145, n=149) | 0.91 | 0.94
  Week 8 (n=132, n=136) | 0.89 | 0.93
  Week 12 (n=119, n=123) | 0.85 | 0.90
  Week 16 (n=102, n=113) | 0.84 | 0.89
  Week 20 (n=102, n=111) | 0.84 | 0.89
  Week 24 (n=91, n=95) | 0.82 | 0.87
  Week 28 (n=79, n=85) | 0.79 | 0.85
  Week 32 (n=74, n=82) | 0.79 | 0.84
  Week 36 (n=74, n=76) | 0.79 | 0.83
  Week 40 (n=74, n=70) | 0.79 | 0.82
  Week 44 (n=74, n=70) | 0.79 | 0.82
  Week 48 (n=74, n=70) | 0.79 | 0.82
  Week 52 (n=19, n=70) | 0.76 | 0.82
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Test type: Superiority or Other; p = 0.381, Log Rank — p-value for equality of survival curves; stratified log-rank test, conrolling for type of index mood episode; Hazard Ratio (HR) = 0.784, 95% CI 2-sided [0.454 to 1.354] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Proportion of Participants Without Discontinuation for Any Reason in the Double-blind Relapse Assessment Phase (Phase 2)
Description: Proportion of Participants without Discontinuation Through Week 52(Kaplan-Meier's estimated survival rate).
Time Frame: Weeks 0, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 1
Measure: Number; unit: Proportion of Participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 173 | 178
Proportion of Participants
  Week 0 (n=173, n=178) | 0.95 | 0.99
  Week 2 (n=164, n=175) | 0.90 | 0.91
  Week 4 (n=155, n=161) | 0.84 | 0.84
  Week 6 (n=145, n=149) | 0.79 | 0.78
  Week 8 (n=135, n=138) | 0.71 | 0.70
  Week 12 (n=122, n=124) | 0.61 | 0.65
  Week 16 (n=103, n=115) | 0.55 | 0.62
  Week 20 (n=95, n=110) | 0.53 | 0.59
  Week 24 (n=90, n=104) | 0.46 | 0.51
  Week 28 (n=78, n=89) | 0.41 | 0.47
  Week 32 (n=70, n=83) | 0.38 | 0.44
  Week 36 (n=64, n=77) | 0.36 | 0.41
  Week 40 (n=61, n=72) | 0.34 | 0.39
  Week 44 (n=57, n=69) | 0.33 | 0.38
  Week 48 (n=56, n=66) | 0.32 | 0.37
  Week 52 (n=19, n=65) | 0.25 | 0.37
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Test type: Superiority or Other; p = 0.295, Log Rank — p-value for equality of survival curves; stratified Log-Rank Test, controlling for type of index mood episode; Hazard Ratio (HR) = 0.871, 95% CI 2-sided [0.672 to 1.128] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Deaths, Treatment-Emergent Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation of Study Medication, Treatment-Emergent AEs and Treatment-Emergent Extrapyramidal Syndrome (EPS)-Related AEs
Description: AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a cancer, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: Throughout Phase 2 (up to 52 weeks)
Population: The Phase 2 Safety Sample comprises all patients who are randomized into Phase 2 and take at least one dose of double-blind medication in Phase 2, as indicated on the study therapy form.
Measure: Number; unit: participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
participants
  Deaths | 0 | 0
  Treatment-Emergent SAEs | 9 | 5
  Suicide-Related SAEs | 0 | 0
  AEs Leading to Discontinuation of Study Medication | 12 | 14
  Treatment-Emergent AEs | 111 | 124
  Treatment-Emergent EPS-Related AEs | 15 | 28

6. Secondary Outcome: Adjusted Mean Change From Baseline in Body Weight, Phase 2
Description: Adjusted for index mood episode and baseline assessment
Time Frame: Baseline, Week 52
Population: Participants from the phase 2 Safety Sample who had body weight evaluation at baseline and week 52 LOCF.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 143 | 151
kg | -1.81 (0.48) | 0.43 (0.47)
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Week 52 LOCF; Test type: Superiority or Other; p = 0.001, ANCOVA — ANOVA (main effects=double-blind treatment, covariate=index mood episode) used for baseline comparisons. ANCOVA (main effects=double-blind treatment, covariates=index mood episode & baseline assessment) used for mean change from baseline comparisons; Treatement Difference = 2.24, 95% CI 2-sided [0.91 to 3.57] — Aripiprazole vs. placebo

7. Secondary Outcome: Number of Participants Showing Clinically Relevant Weight Loss by Study Week
Description: Weight Loss of at least a 7% decrease from Baseline.
Time Frame: Weeks 12, 24, 36, 52
Population: Observed cases (OC) data set (actual observation at each visit), Last observation carried forward (LOCF) data set (data recorded at a given visit or, if no observation is recorded at that visit, data carried forward from the previous visit), and Overall, Phase 2 Safety Sample; n=number assessed at given time point.
Measure: Number; unit: Participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
Participants
  Week 12 (n=105, 107) | 7 | 9
  Week 24 (n=84, 87) | 8 | 9
  Week 36 (n=54, 67) | 10 | 6
  Week 52 (n=49, 56) | 10 | 6
  Week 52 LOCF (n=143, 151) | 22 | 13
  At Any Time (n=147, 154) | 26 | 19
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Week 52 LOCF; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.56, 95% CI 2-sided [0.29 to 1.07] — aripiprazole/placebo
Statistical Analysis 2: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; At Any Time; Test type: Superiority or Other; p = 0.194, Cochran-Mantel-Haenszel

8. Secondary Outcome: Number of Participants Showing Clinically Relevant Weight Gain by Study Week
Description: Weight gain of at least a 7% increase from Baseline.
Time Frame: Weeks 12, 24, 36, 52
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
Participants
  Week 12 (n=105, 107) | 2 | 4
  Week 24 (n=84, 87) | 3 | 10
  Week 36 (n=54, 67) | 5 | 14
  Week 52 (n=49, 56) | 2 | 7
  Week 52 LOCF (n=143, 151) | 5 | 18
  At Any Time (n=147, 154) | 8 | 27
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Week 52 LOCF; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; relative risk = 3.41, 95% CI 2-sided [1.30 to 8.94]
Statistical Analysis 2: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

9. Secondary Outcome: Adjusted Mean Change From Baseline in BMI by Study Week
Description: Adjusted for index mood episode and baseline assessment.
Time Frame: Baseline, Weeks 12, 24, 36, 52
Population: as for outcome 7
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
kg/m2
  Baseline (n=143, 150) | 30.77 (0.63) | 30.13 (0.61)
  Change from Baseline Week 12 (n=105, 107) | -0.39 (0.15) | -0.03 (0.15)
  Change from Baseline Week 24 (n=84, 87) | -0.60 (0.20) | 0.14 (0.20)
  Change from Baseline Week 36 (n=54, 67) | -0.63 (0.33) | 0.34 (0.30)
  Change from Baseline Week 52 (n=49, 56) | -0.73 (0.37) | 0.19 (0.34)
  Change from Baseline Week 52 LOCF (n=143, 150) | -0.62 (0.17) | 0.17 (0.17)
  Highest Change from Baseline (n=143, 150) | -0.02 (0.15) | 0.61 (0.14)
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Baseline; Test type: Superiority or Other; p = 0.467, ANCOVA — Means, treatment differences between aripiprazole and placebo, 95% confidence intervals for the differences and the p-values for treatment comparisons are based on ANOVA/ANCOVA model; ANCOVA model, with double-blind treatment as main effects and index mood episode as covariate, is used for Baseline comparisons; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-2.37 to 1.09] — aripiprazole - placebo
Statistical Analysis 2: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at Week 12; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; ANCOVA (main effects=double-blind treatment, covariates=index mood episode & baseline assessment) used for mean change from baseline comparisons; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-0.06 to 0.78] — aripiprazole - placebo
Statistical Analysis 3: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 24; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 9, analysis 2]; Mean Difference (Final Values) = 0.75, 95% CI 2-sided [0.19 to 1.30] — aripiprazole - placebo
Statistical Analysis 4: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 36; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 9, analysis 2]; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [0.08 to 1.86] — aripiprazole - placebo
Statistical Analysis 5: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 52; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 9, analysis 2]; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-0.08 to 1.92] — aripiprazole - placebo
Statistical Analysis 6: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 9, analysis 2]; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [0.31 to 1.26] — aripiprazole - placebo
Statistical Analysis 7: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Highest Change from baseline; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 9, analysis 2]; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [0.23 to 1.04] — aripiprazole - placebo

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities Occurring During Double-Blind Treatment
Description: Abbreviations and further description used in table: Sinus tachycardia, ≥120 beats per minute (bpm) and ↑ ≥15 bpm & no current diagnosis of supraventricular or ventricular tachycardia/atrial fibrillation (AF)/atrial flutter/ other rhythm abnormality. Sinus bradycardia, ≤ 50 bpm and ↓ 15 bpm & no current diagnosis of AF/atrial flutter/other rhythm abnormality. Supraventricular premature beat (SPB), Ventricular premature beat (VPB), Atroventricular (A-V). Other intraventricular block, QRS ≥0.12 sec and ↑ ≥0.02 sec & no current diagnosis of left or right bundle branch block.
Time Frame: Throughout the study, up to Week 52
Population: Participants with ECG evaluation from the phase 2 Safety Sample (all patients who are randomized into Phase 2 and take at least one dose of double-blind medication in Phase 2, as indicated on the study therapy form.)
Measure: Number; unit: particiapnts
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 124 | 132
particiapnts
  Tachycardia: ≥ 120 bpm and ↑ ≥ 15 bpm | 1 | 1
  Bradycardia: ≤ 50 bpm and ↓ 15 bpm | 2 | 0
  Sinus Tachycardia: ≥ 120 bpm and ↑ ≥ 15 bpm | 1 | 0
  Sinus Bradycardia: ≤ 50 bpm and ↓ 15 bpm | 2 | 0
  SPB: not present → present (see description) | 0 | 0
  VPB: not present → present (see description) | 2 | 1
  Supraventricular Tachycardia: not present→ present | 0 | 0
  Ventricular Tachycardia: not present → present | 0 | 0
  Atrial Fibrillation (AF): not present → present | 0 | 0
  AF With Rapid Ventricular Response | 0 | 0
  Atrial Flutter: not present → present | 0 | 1
  1st Degree A-V Block: PR ≥0.20 sec and ↑ ≥0.05 sec | 0 | 0
  2nd Degree A-V Block: not present → present | 0 | 0
  3rd Degree A-V Block: not present → present | 0 | 0
  Left Bundle Branch Block: not present → present | 0 | 0
  Right Bundle Branch Block: not present → present | 6 | 4
  Pre-excitation Syndrome: not present → present | 0 | 0
  Other Intraventricular Conduction: see description | 0 | 0
  Acute Infarction: not present → present | 0 | 0
  Subacute (recent) Infarction: not present→ present | 0 | 0
  Old Infarction: not present → present | 1 | 0
  Myocardial Ischemia: not present → present | 0 | 0
  Symmetrical T-Wave Inversions: not present→present | 0 | 0
  QTc Bazett: > 450 msec | 5 | 6
  QTc (.37): > 450 msec | 0 | 0
  QTc (.33): > 450 msec | 0 | 1

11. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Vital Sign Abnormalities Occurring During Double-Blind Treatment
Description: In order to be identified as clinically relevant abnormal, an on-drug value must meet the Criterion Value (CV) and also represent a change from the patient's pretreatment value of at least the Change Relative to Baseline (CRB) magnitude. Heart Rate CV: 120 beats per minute (bpm), CRB: increase of ≥15 / CV: 50 bpm, CRB: decrease of ≥15. Systolic BP CV: 180 mmHg, CRB: increase of ≥20 / CV: 90 mmHg, CRB: decrease of ≥20. Diastolic BP CV: 105 mmHg, CRB: increase of ≥15 / CV: 50 mmHg, CRB: decrease of ≥15.
Time Frame: Up to 52 Weeks
Population: Phase 2 Safety Sample (all patients who are randomized into Phase 2 and take at least one dose of double-blind medication in Phase 2, as indicated on the study therapy form).
Measure: Number; unit: participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
participants
  Systolic BP, supine-Increase (n=160,168) | 3 | 1
  Systolic BP, supine-Decrease (n=160,168) | 7 | 5
  Systolic BP, standing-Increase (n=153, 157) | 3 | 0
  Systolic BP, standing-Decrease (n=153,157) | 2 | 4
  Diastolic BP, supine-Increase (n=160,168) | 2 | 0
  Diastolic BP, supine-Decrease (n=160,168) | 0 | 3
  Diastolic BP, standing-Increase (n=153,157) | 6 | 1
  Diastolic BP, standing-Decrease (n=153,157) | 0 | 1
  Heart Rate, supine-Increase (n=160,168) | 0 | 0
  Heart Rate, supine-Decrease (n=160,168) | 3 | 0
  Heart Rate, standing-Increase (n=153, 157) | 4 | 2
  Heart Rate, standing-Decrease (n=153, 157) | 1 | 0

12. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Abnormalities Occurring During Double-Blind Treatment (Phase 2)
Description: Chemistry, hematology, and urinalysis abnormalities.Abbreviations used: alanine aminotransferase (ALT), institutional upper limit of normal (ULN), aspartate aminotransferase (AST), alkaline phosphatase (ALP), lactate dehydrogenase (LDH), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), baseline (BL)
Time Frame: Throughout Phase 2 of the study, up to Week 52
Population: Phase 2 safety sample
Measure: Number; unit: particiapnts
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
particiapnts
  ALT ≥3 x ULN (n=151,157) | 3 | 0
  AST ≥3 x ULN (n=151, 157) | 2 | 1
  ALP ≥3 x ULN (n=151, 157) | 0 | 0
  LDH ≥3 x ULN (n=151, 158) | 0 | 0
  BUN ≥30 mg/dL (n=151, 158) | 0 | 2
  Creatine kinase (n=3, 1) | 0 | 0
  Creatinine ≥2.0 mg/dL (n=151, 157) | 0 | 0
  Uric acid (n=151, 157) | 0 | 2
  Bilirubin (total) ≥ 2.0 mg/dL (n=152, 157) | 0 | 0
  Prolactin (n=152, 158) | 32 | 18
  Cholesterol Total (n=151, 157) | 22 | 28
  Cholesterol Total (fasting) (n=126, 124) | 17 | 25
  Cholesterol Total (non-fasting) (n=68, 75) | 9 | 7
  Glucose Fasting Serum (n=126, 125) | 15 | 13
  HDL-C (n=151, 158) | 53 | 38
  HDL-C (fasting) (n=126, 125) | 44 | 25
  HDL-C (non-fasting) (n=68, 75) | 23 | 19
  LDL-C (n=151, 157) | 17 | 26
  LDL-C (fasting) (n=126, 124) | 14 | 22
  LDL-C (non-fasting) (n=68, 75) | 7 | 5
  Triglycerides (n=151, 157) | 0 | 0
  Triglycerides (fasting) (n=126, 124) | 26 | 29
  Triglycerides (non-fasting) (n=68, 75) | 19 | 20
  Sodium serum (n=152, 158) | 1 | 0
  Potassium serum (n=152, 158) | 0 | 0
  Chloride serum (n=152, 158) | 0 | 0
  Calcium (n=151, 157) | 0 | 0
  Hemoglobin ≤11.5 g/dL(m)/≤9.5 g/dL(f) (n=152, 156) | 1 | 0
  Hematocrit ≤37(m)/≤32(f) & 3 ↓from BL (n=152,156) | 1 | 3
  Leukocytes ≤2800 mm^3 or ≥16000 mm^3 (n=152, 156) | 0 | 2
  Eosinophils relative (calculated)≥10% (n=152, 156) | 2 | 2
  Neutrophils relative (calculated)≤15% (n=152, 156) | 0 | 0
  Platelets ≤75,000 mm3 or ≥700,000 mm3 (n=152,155) | 0 | 0
  Protein urine increase of ≥2 units (n=145, 152) | 0 | 0
  Glucose urine (n=149, 155) | 0 | 0

13. Secondary Outcome: Summary of Concomitant Medications, Phase 1
Time Frame: Phase 1 (9 to 24 Week Single-blind Stabilization Phase)
Population: Phase 1 Safety Sample (all patients who take at least one dose of singleblind aripiprazole in Phase 1, as indicated on the study therapy form).
Measure: Number; unit: participants
Arm/Group | Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole
Number analyzed (Participants) | 787
participants
  Any central nervous system Medication | 550
  Analgesic | 2
  Anesthetic, general | 1
  Anesthetic, local | 3
  Anticholinergic | 98
  Antidepressant | 12
  Antiepileptic | 48
  Antimigraine prep | 12
  Antipsychotic | 20
  Anxiolytic | 267
  Hypnotic & Sedative | 206
  Opiod | 78
  Other Analgesic & Antipyretic | 253
  Other Nervous System Drug | 1
  Psychostimulant | 2
  Any extrapyramidal syndrome Medication | 98
  Benztropine | 98

14. Secondary Outcome: Summary of Concomitant Medications, Phase 2
Time Frame: Phase 2 (52 Week Double-blind Relapse Assessment Phase)
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
participants
  Any central nervous system Medication | 120 | 132
  Anesthetic, local | 1 | 0
  Anticholinergic | 21 | 25
  Antidepressant | 3 | 1
  Antiepileptic | 8 | 11
  Antimigraine prep | 1 | 3
  Antipsychotic | 5 | 3
  Anxiolytic | 63 | 62
  Hypnotic & Sedative | 50 | 41
  Opiod | 20 | 14
  Other Analgesic & Antipyretic | 53 | 66
  Psychostimulant | 0 | 1
  Any extrapyramidal syndrome Medication | 25 | 35
  Benztropine | 25 | 35
  Trihexyphenidyl | 1 | 1

15. Secondary Outcome: Adjusted Mean Change From Baseline in Simpson-Angus Scale (SAS) Total Score
Description: The SAS is a 10-item instrument used to evaluate the presence and severity of parkinsonian symptomatology. The ten items focus on rigidity rather than bradykinesia, and do not assess subjective rigidity or slowness. Items are rated for severity on a 0-4 scale, with definitions given for each anchor point. The total SAS Score has a possible range from 10 to 50. Negative change scores indicate improvement.
Time Frame: Baseline, Weeks 8, 24, 36, 52
Population: Observed cases (OC) data set (actual observation at each visit), Last observation carried forward (LOCF) data set (data recorded at a given visit or, if no observation is recorded at that visit, data carried forward from the previous visit). n=number of participants analyzed at timepoint.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
units on a scale
  Baseline (n=125, 128) | 10.59 (0.12) | 10.58 (0.12)
  Change from Baseline at Week 8 (n=125, 124) | -0.20 (0.10) | 0.05 (0.10)
  Change from Baseline at Week 24 (n=85, 89) | -0.21 (0.13) | 0.03 (0.13)
  Change from Baseline at Week 36 (n=54, 67) | -0.38 (0.11) | -0.14 (0.10)
  Change from Baseline at Week 52 (n=50, 56) | -0.35 (0.13) | -0.05 (0.12)
  Change from Baseline at Week 52 LOCF (n=152, 161) | -0.22 (0.10) | 0.02 (0.10)
  Highest Change from Baseline (n=152, 161) | 0.03 (0.12) | 0.34 (0.11)
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Baseline; Test type: Superiority or Other; p = 0.971, ANOVA — [p-value comment as in outcome 9, analysis 1]; ANOVA model, with double-blind treatment as main effects, is used for Baseline comparisons; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.35 to 0.34] — aripiprazole - placebo
Statistical Analysis 2: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 8; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; ANCOVA (main effects=double-blind treatment, covariate=baseline assessment) used for mean change from baseline comparisons; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.03 to 0.51] — aripiprazole - placebo
Statistical Analysis 3: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 24; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.13 to 0.60] — aripiprazole - placebo
Statistical Analysis 4: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at Week 36; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.06 to 0.55] — aripiprazole - placebo
Statistical Analysis 5: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 52; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.06 to 0.65] — aripiprazole - placebo
Statistical Analysis 6: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.095, ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.04 to 0.52] — aripiprazole - placebo
Statistical Analysis 7: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Highest change from Baseline; Test type: Superiority or Other; p = 0.061, ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-0.01 to 0.63] — aripirazole - placebo

16. Secondary Outcome: Adjusted Mean Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS is an assessment of movement dysfunctions. It is a 12-item instrument assessing abnormal involuntary movements associated with antipsychotic drugs and 'spontaneous' motor disturbance related to the illness itself. Scoring the AIMS consists of rating the severity of movement in 3 main anatomic areas (facial/oral, extremities, and trunk), based on a five-point scale (0=none, 4=severe). The AIMS Total Score has a possible range from 0 to 28. Negative change scores indicate improvement in movement dysfunction.
Time Frame: Baseline, Weeks 8, 24, 36, 52
Population: as for outcome 15
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
units on a scale
  Baseline (n=125, 128) | 0.21 (0.07) | 0.14 (0.07)
  Change from Baseline at Week 8 (n=124, 124) | -0.05 (0.05) | 0.06 (0.06)
  Change from Baseline at Week 24 (n=85, 89) | -0.01 (0.06) | 0.04 (0.05)
  Change from Baseline at Week 36 (n=54, 67) | -0.09 (0.08) | 0.13 (0.07)
  Change from Baseline at Week 52 (n=50, 56) | -0.11 (0.04) | -0.05 (0.04)
  Change from Baseline at Week 52 LOCF (n=153, 161) | 0.05 (0.06) | -0.01 (0.06)
  Highest Change from Baseline (n=153, 161) | 0.10 (0.07) | 0.14 (0.07)
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Baseline; Test type: Superiority or Other; p = 0.458, ANOVA — [p-value comment as in outcome 9, analysis 1]; ANOVA model, controlling for treatment, is used for baseline estimates; Mean Difference (Final Values) = -0.07, 95% CI [-0.25 to 0.11] — aripiprazole - placebo
Statistical Analysis 2: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at Week 8; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.05 to 0.26] — aripiprazole - placebo
Statistical Analysis 3: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 24; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.11 to 0.20] — aripiprazole - placebo
Statistical Analysis 4: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at Week 36; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [0.00 to 0.42] — aripiprazole - placebo
Statistical Analysis 5: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at week 52; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.05 to 0.16] — aripiprazole - placebo
Statistical Analysis 6: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.515, ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.22 to 0.11] — aripiprazole - placebo
Statistical Analysis 7: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Highest Change from Baseline; Test type: Superiority or Other; p = 0.730, ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.16 to 0.23] — aripiprazole - placebo

17. Secondary Outcome: Adjusted Mean Change From Baseline in Barnes Akathisia Global Clinical Assessment,
Description: The Barnes Akathisia Rating Scale is a 4-item scale to assess presence and severity of drug-induced akathisia, including both objective items and subjective items, together with a global clinical assessment of akathisia. Global assessment is made on a scale of 0 to 5 with comprehensive definitions provided for each anchor point on scale: 0=absent; 1=questionable; 2=mild akathisia; 3=moderate akathisia; 4=marked akathisia; 5=severe akathisia. Score has a possible range from 0 (absent) to 5 (severe akathisia). Negative change scores indicate improvement in akathisia.
Time Frame: Baseline, Weeks 8, 24, 36, 52
Population: as for outcome 15
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Number analyzed (Participants) | 165 | 176
units on a scale
  Baseline (n=125, 128) | 0.22 (0.05) | 0.27 (0.05)
  Change from Baseline at Week 8 (n=125, 124) | -0.12 (0.05) | 0.04 (0.05)
  Change from Baseline at Week 24 (n=85, 89) | -0.09 (0.05) | -0.06 (0.05)
  Change from Baseline at Week 36 (n=54, 67) | -0.18 (0.05) | -0.18 (0.04)
  Change from Baseline at Week 52 (n=50, 56) | -0.20 (0.04) | -0.17 (0.04)
  Change from Baseline at Week 52 LOCF (n=153, 161) | -0.11 (0.04) | -0.05 (0.04)
  Highest Change from Baseline (n=153, 161) | -0.02 (0.05) | 0.15 (0.05)
Statistical Analysis 1: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Baseline; Test type: Superiority or Other; p = 0.435, ANOVA — Means, mean differences, 95% confidence intervals for the differences, and the p-values are based on ANOVA/ANCOVA model; ANOVA, controlling for treatment, used for baseline estimates; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.08 to 0.20] — aripiprazole - placebo
Statistical Analysis 2: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at Week 8; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.04 to 0.30] — aripiprazole - placebo
Statistical Analysis 3: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at Week 24; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.11 to 0.17] — aripiprazole - placebo
Statistical Analysis 4: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 36; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.13 to 0.13] — aripiprazole - placebo
Statistical Analysis 5: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from baseline at Week 52; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.08 to 0.14] — aripiprazole - placebo
Statistical Analysis 6: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.358, ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.06 to 0.17] — aripiprazole - placebo
Statistical Analysis 7: Comparison: Phase 2 Double-Blind Treatment: Lamotrigine + Placebo vs Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole; Highest Change from Baseline; Test type: Superiority or Other; p = 0.021, ANCOVA — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 15, analysis 2]; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.03 to 0.31] — aripiprazole - placebo

ADVERSE EVENTS:
Arm/Group | Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole
Serious Adverse Events (participants affected / at risk) | 32/787 | 9/165 | 5/176
Other Adverse Events (participants affected / at risk) | 545/787 | 61/165 | 74/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole (N=787) | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo (N=165) | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole (N=176)
CARDIAC DISORDER (Cardiac disorders) | 0 | 0 | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 1 | 0
WOLFF-PARKINSON-WHITE SYNDROME (Cardiac disorders) | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0
PHYSICAL ASSAULT (Social circumstances) | 1 | 0 | 0
MANIA (Psychiatric disorders) | 3 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 0
AGITATION (Psychiatric disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 3 | 0 | 1
PANIC ATTACK (Psychiatric disorders) | 1 | 0 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 2 | 0 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 8 | 0 | 0
BIPOLAR I DISORDER (Psychiatric disorders) | 2 | 2 | 1
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 2 | 0 | 0
HOMICIDAL IDEATION (Psychiatric disorders) | 2 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 1
AKATHISIA (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0 | 0
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0
OBESITY (Metabolism and nutrition disorders) | 0 | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
MENSTRUAL DISORDER (Reproductive system and breast disorders) | 1 | 0 | 0
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 1 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
CHEST PAIN (General disorders) | 3 | 2 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0
VULVAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Single-Blind Treatment, Lamotrigine + Aripiprazole (N=787) | Phase 2 Double-Blind Treatment: Lamotrigine + Placebo (N=165) | Phase 2 Double-Blind Treatment: Lamotrigine + Aripiprazole (N=176)
ANXIETY (Psychiatric disorders) | 73 | 6 | 13
INSOMNIA (Psychiatric disorders) | 138 | 19 | 13
AGITATION (Psychiatric disorders) | 65 | 8 | 11
RESTLESSNESS (Psychiatric disorders) | 55 | 2 | 3
HEADACHE (Nervous system disorders) | 92 | 13 | 8
SEDATION (Nervous system disorders) | 62 | 3 | 1
AKATHISIA (Nervous system disorders) | 196 | 10 | 19
DIZZINESS (Nervous system disorders) | 40 | 3 | 2
SOMNOLENCE (Nervous system disorders) | 42 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 103 | 6 | 7
VOMITING (Gastrointestinal disorders) | 40 | 1 | 1
DRY MOUTH (Gastrointestinal disorders) | 44 | 3 | 4
URINARY TRACT INFECTION (Infections and infestations) | 35 | 9 | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 34 | 13 | 12
BACK PAIN (Musculoskeletal and connective tissue disorders) | 26 | 5 | 9
FATIGUE (General disorders) | 74 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.